CLINICAL TRIAL: NCT02217462
Title: Diet, Obesity, and Weight Change in Pregnancy
Brief Title: Pregnancy Eating Attributes Study
Acronym: PEAS
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of North Carolina, Chapel Hill (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HHSN275201300015C
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy
Keywords: pregnancy; gestational weight gain; dietary intake; food reward
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma White and red blood cells Urine Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women

SUMMARY:
The primary purpose of this observational cohort study is to examine the role of "food reward" in maternal diet and weight change during pregnancy and postpartum. The study will further examine the importance of food reward in the context of behavioral control and other related aspects of eating behavior, as well as weight-related biomedical, psychosocial and behavioral factors including genetics, physical activity, stress, sleep and depression. Four hundred and fifty women of varying baseline weight status will be enrolled early in pregnancy (before 12 weeks postpartum) and followed until 1 year postpartum. Assessments will occur at baseline (<12 weeks postpartum), during pregnancy at 13-18 weeks gestation, 16-22 weeks, and 28-32 weeks, and postpartum at 4-6 weeks, 6 months, 9 months and 12 months. Measures will include assessments of food reward and related constructs, dietary intake, other health behaviors, and anthropometrics. Clinical data and biological specimens will be obtained. Infant anthropometrics and feeding practices will also be assessed. Primary exposures include aspects of food reward and behavioral control, which will be assessed in multiple ways to maximize information and utility. Primary outcomes include gestational weight gain, postpartum weight retention and dietary quality.

ELIGIBILITY:
Inclusion Criteria:

* Female confirmed pregnant <12 weeks at screening
* Uncomplicated singleton pregnancy anticipated
* Age >=18 and <45 at screening
* Willingness to undergo study procedures and provide informed consent for her participation and assent for the baby's participation
* BMI >=18.5 (to qualify as normal: 18.5-24.9; overweight 25-29.9; or obese : >=30)
* Able to complete self-reported assessments in English
* Access to Internet with email to complete self-reported assessments
* Plan to deliver at UNC Hospital
* Plan to remain in the area for 1 year following delivery

Exclusion Criteria:

* Pre-existing diabetes (type 1 or type 2)
* Multiple pregnancy
* Participant-reported eating disorder
* Any fetal anomaly requiring surgery with hospital admission following delivery (e.g. NTDs, gastroschisis, cardiac defects, Trisomy 21)
* Any medical condition contraindicating participation in the study such as chronic illnesses or use of medication that could affect diet or weight e.g. cancer, HIV, active renal disease, MI in the last 6 months, chronic steroid use, thyroid disease requiring medication, or autoimmune disease (rheumatoid arthritis, lupus, antiphospholipid antibody syndrome, scleroderma)
* Psychosocial condition contraindicating participation in the study such as bipolar, schizophrenia, major affective disorder, substance abuse.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: PEAS is a prospective observational study of N=450 women without evidence of psychiatric or eating disorders, recruited in early pregnancy (≤12 weeks), targeting N=150 in each weight status group: normal weight (BMI 18.5-24.9), overweight (BMI 25-29.9) and obese (BMI >=30). Women will be followed through pregnancy and until 1 year postpartum, along with their infants from birth to 1 year, with collection of blood, stool, and urine specimens, previous and current medical information, dietary intake and eating behaviors, anthropometrics, and demographic information.
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Body weight | <12 weeks pregnancy; 16-22 weeks pregnancy; 28-32 weeks pregnancy; delivery; 4-6 weeks postpartum; 6 months postpartum; 1 year postpartum
Dietary intake | <12 weeks pregnancy; 16-22 weeks pregnancy; 28-32 weeks pregnancy; 4-6 weeks postpartum; 6 months postpartum; 1 year postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Tonja R. Nansel, PhD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- UNC Hospitals Obstetrics Clinic; Timberlylne Obstetrics & Gynecology Clinic, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Lipsky LM, Burger KS, Faith MS, Shearrer GE, Nansel TR. Eating in the absence of hunger is not associated with weight, self-reported eating behaviors, or well-being in pregnant adults: Prospective cohort study. PLoS One. 2025 Jun 24;20(6):e0325478. doi: 10.1371/journal.pone.0325478. eCollection 2025. PMID 40554514
- [Derived] Cummings JR, Faith MS, Lipsky LM, Liu A, Mooney JT, Nansel TR. Prospective relations of maternal reward-related eating, pregnancy ultra-processed food intake and weight indicators, and feeding mode with infant appetitive traits. Int J Behav Nutr Phys Act. 2022 Aug 3;19(1):100. doi: 10.1186/s12966-022-01334-9. PMID 35922793
- [Derived] Cummings JR, Lipsky LM, Schwedhelm C, Liu A, Nansel TR. Associations of ultra-processed food intake with maternal weight change and cardiometabolic health and infant growth. Int J Behav Nutr Phys Act. 2022 May 26;19(1):61. doi: 10.1186/s12966-022-01298-w. PMID 35619114
- [Derived] Temmen CD, Lipsky LM, Faith MS, Nansel TR. Prospective relations between maternal emotional eating, feeding to soothe, and infant appetitive behaviors. Int J Behav Nutr Phys Act. 2021 Aug 11;18(1):105. doi: 10.1186/s12966-021-01176-x. PMID 34380499
- [Derived] Schwedhelm C, Lipsky LM, Shearrer GE, Betts GM, Liu A, Iqbal K, Faith MS, Nansel TR. Using food network analysis to understand meal patterns in pregnant women with high and low diet quality. Int J Behav Nutr Phys Act. 2021 Jul 23;18(1):101. doi: 10.1186/s12966-021-01172-1. PMID 34301273
- [Derived] Betts GM, Lipsky LM, Temmen CD, Siega-Riz AM, Faith MS, Nansel TR. Poorer mental health and sleep quality are associated with greater self-reported reward-related eating during pregnancy and postpartum: an observational cohort study. Int J Behav Nutr Phys Act. 2021 May 1;18(1):58. doi: 10.1186/s12966-021-01124-9. PMID 33933087
- [Derived] Nansel TR, Lipsky LM, Faith M, Liu A, Siega-Riz AM. The accelerator, the brake, and the terrain: associations of reward-related eating, self-regulation, and the home food environment with diet quality during pregnancy and postpartum in the pregnancy eating attributes study (PEAS) cohort. Int J Behav Nutr Phys Act. 2020 Nov 23;17(1):149. doi: 10.1186/s12966-020-01047-x. PMID 33228724
- [Derived] Lipsky LM, Burger KS, Faith MS, Shearrer GE, Nansel TR. Eating in the Absence of Hunger Is Related to Worse Diet Quality throughout Pregnancy. J Acad Nutr Diet. 2021 Mar;121(3):501-506. doi: 10.1016/j.jand.2020.09.037. Epub 2020 Nov 3. PMID 33158801
- [Derived] Lipsky LM, Burger KS, Faith MS, Siega-Riz AM, Liu A, Shearrer GE, Nansel TR. Pregnant Women Consume a Similar Proportion of Highly vs Minimally Processed Foods in the Absence of Hunger, Leading to Large Differences in Energy Intake. J Acad Nutr Diet. 2021 Mar;121(3):446-457. doi: 10.1016/j.jand.2020.09.036. Epub 2020 Oct 24. PMID 33109504
- [Derived] Hill C, Lipsky LM, Betts GM, Siega-Riz AM, Nansel TR. A Prospective Study of the Relationship of Sleep Quality and Duration with Gestational Weight Gain and Fat Gain. J Womens Health (Larchmt). 2021 Mar;30(3):405-411. doi: 10.1089/jwh.2020.8306. Epub 2020 Sep 18. PMID 32945728
- [Derived] Nansel TR, Lipsky LM, Siega-Riz AM, Burger K, Faith M, Liu A. Pregnancy eating attributes study (PEAS): a cohort study examining behavioral and environmental influences on diet and weight change in pregnancy and postpartum. BMC Nutr. 2016;2:45. doi: 10.1186/s40795-016-0083-5. Epub 2016 Jul 15. PMID 28663822